CLINICAL TRIAL: NCT00888823
Title: Multicentre, Phase I/II Study of Fractionated Stereotactic Radiotherapy for Medically Inoperable Early Stage Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Phase I/II Study of Fractionated Stereotactic Radiotherapy for Early Stage Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24541/ethics24761
Record Dates: First submitted 2009-04-27; First posted 2009-04-28 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Fractionated stereotactic radiotherapy; Medically inoperable; Image-guided radiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: Stereotactic Radiotherapy — Stereotactic Radiotherapy

SUMMARY:
A new type of treatment called stereotactic radiotherapy has recently been developed in hopes of improving the success of the treatment and improving the convenience to patients, while reducing the side effects. This study is developing stereotactic radiotherapy as a state-of-the-art treatment for lung cancer patients.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary Objectives

* To determine the efficacy of hypofractionated, image guided radiotherapy in treating patients with lung tumours, with the primary outcome being local control at one year.
* To determine the toxicity of high dose, small field,hypofractionated radiotherapy to the lung, based on the RTOG and CTCAE scales.

ELIGIBILITY:
Inclusion Criteria:

* T1-T3N0 non-small cell lung cancer (maximum dimensions of 5cm, T3 by chestwall involvement only)
* Medically inoperable due to co-morbid conditions or patient preference for radiation
* adequate pulmonary function to withstand radical treatment (ie. FEV1 greater than 40% of predicted), as assessed by consulting radiation oncologist
* age greater than or equal to 18, and Karnofsky performance status greater than of equal to 70

Exclusion Criteria:

* Presence of mediastinal metastases or distant metastases
* Life expectancy less than 1 year due to other co-morbid conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-03; Primary Completion 2014-02 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Local Control | One Year

SECONDARY OUTCOMES:
Toxicity | One Year
Quality of Life | One Year

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Tom Baker Cancer Center, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta